CLINICAL TRIAL: NCT00913003
Title: Analgesic Effect of Perioperative Systemic Lidocaine in Patients Undergoing Unilateral Mastectomy Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI terminated employment with the University
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christian Altman, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU0008753
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Pain
Keywords: Lidocaine; Mastectomy; Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Group B using saline as a placebo.
  Interventions: Drug: Placebo
- Lidocaine (Active Comparator): Group A lidocaine infusion and bolus.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine bolus infusion 1.5 mg/kg IV using participants IBW(Ideal Body Weight) Lidocaine infusion after bolus and continuing until 1 hour after skin closure 33.3 mcg/kg/mn IV (IBW)
  Other Names: Group A
  Arms: Lidocaine
Drug: Placebo — Placebo (normal saline) bolus similar to the lidocaine infusion minus active drug
  Other Names: Group B
  Arms: Placebo

SUMMARY:
The aim of this study is to determine if perioperative systemic lidocaine administration will decrease the amount of opioid analgesics required in women undergoing mastectomy surgery. In addition, patients receiving systemic lidocaine will have a lower incidence of post-mastectomy pain syndrome.

This study will have 2 groups. Participants will be randomized into one of each group. The first group will be administered the drug lidocaine prior to surgery and the second group Group B will be administered saline (salt water). This is a blinded study which means the participant will not know which group they have been assigned. The subjects participation will last 12 months (surveys post operatively).

DETAILED DESCRIPTION:
Patients will be recruited up to 21 days prior to the day of surgery. The consent form will be reviewed with the patient, and the patient will be allowed to take a copy home. If the patient does not have an EKG within the past 6 weeks in her medical record, an EKG will be obtained at the time of recruitment. At the time of recruitment, the patient will be randomized using a computer-generated code. Group A will receive lidocaine during surgery, and Group B will receive saline (placebo) during surgery.The study drug will be prepared by the investigator(s). The anesthesiologist and research nurse will be blinded. If necessary in the event of an emergency, these individuals may be unblinded.

Group A (Lidocaine):

Induction: 1.5 mg/kg IV (IBW) bolus, administered prior to Propofol. The maximum loading dose administered will not exceed 150 mg IV Infusion: 33.3 mcg/kg/min IV (IBW), initiated before surgical incision.Discontinue infusion 1 hour after skin closure complete.No other local anesthetics administered intra-operatively

Group B (Saline):

Induction: IV bolus, administered prior to Propofol Infusion: Initiate before surgical incision (rate calculated as if for lidocaine infusion). Discontinue infusion 1 hour after skin closure complete No local anesthetics administered intra-operatively. Baseline thermal quantitative sensory testing (QST) scores will be obtained pre-operatively using TSA-II Neuro Sensory Analyzer (Medoc Advanced Medical Systems, Durham, NC).

Baseline Modified Quality of Recovery (MQoR-40) Survey will be obtained on the morning of surgery.

Preoperative anxiety, depression, and pain characterization will be measured within 24 hours of the time of surgery using a validated questionnaire (Hospital Anxiety and Depression Scale). If the questionnaire responses indicate the patient is experiencing depressive symptoms, the patient will be notified of the results and instructed to follow up with her primary care physician.

Intraoperatively, patients will receive a standardized anesthetic (management protocol attached).

Two blood samples for lidocaine levels will be obtained on subjects. The first lidocaine blood sample will be collected after the lidocaine/placebo bolus in the operating room. The second lidocaine blood sample will be obtained when the lidocaine/placebo infusion has been discontinued (one hour after skin closure). A total of 5 mLs of blood will be obtained.

Patients will be examined daily by a research nurse while admitted to the hospital. Daily pain scores will be noted, as will complications related to the perioperative period. If the subject is discharged within 24 hours the research nurse will call by phone to ask the subject about pain 0-10 and type and amount of pain relievers used since discharge.MQoR-40 will be administered on the day of discharge. It will be repeated at 6 weeks, 6 months, and 12 months after surgery. Patients will complete the Mastectomy Patient Follow-Up, Modified LANNS Pain Scale, and McGill Pain questionnaires at 6 months and 12 months after surgery for detection of Post-Mastectomy Pain Syndrome (PMPS).

The definition of PMPS will be: The presence of a dull, burning,and aching sensation in the anterior chest, arm, and axilla exacerbated by movement of the shoulder girdle.

Appendix 1-Anesthetic Management Protocol Appendix 2-HADS Appendix 3-MQoR-40 Appendix 4-Modified LANNS and McGill Appendix 5-Follow-Up Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Gender: Female
* ASA Physical Status I-III
* Non-pregnant
* Surgery: Unilateral total or segmental mastectomy
* Language: English speaking
* Consent: Obtained

Exclusion Criteria:

* Age: Under 18 or over 65 years
* ASA Physical Status >III
* Pregnancy
* Language: Non-English speaking
* Allergy to Lidocaine or amide local anesthetics
* Contraindication to succinylcholine
* History and/or EKG evidence of conduction defect
* Renal failure (Creatinine >1.7 mg/dL)
* Patient expected to remain intubated after procedure
* Chronic home opioid or steroid use
* Opioid use within one week prior to procedure
* Drug or alcohol abuse
* Inability to use PCA

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Altman, M.D., Principal Investigator — Northwestern University

REFERENCES:
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Joshi GP. Multimodal analgesia techniques and postoperative rehabilitation. Anesthesiol Clin North Am. 2005 Mar;23(1):185-202. doi: 10.1016/j.atc.2004.11.010. PMID 15763418
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Background] Macdonald L, Bruce J, Scott NW, Smith WC, Chambers WA. Long-term follow-up of breast cancer survivors with post-mastectomy pain syndrome. Br J Cancer. 2005 Jan 31;92(2):225-30. doi: 10.1038/sj.bjc.6602304. PMID 15655557
- [Background] McCleane G. Intravenous lidocaine: an outdated or underutilized treatment for pain? J Palliat Med. 2007 Jun;10(3):798-805. doi: 10.1089/jpm.2006.0209. PMID 17592992
- [Background] Owczuk R, Wujtewicz MA, Sawicka W, Piankowski A, Polak-Krzeminska A, Morzuch E, Wujtewicz M. The effect of intravenous lidocaine on QT changes during tracheal intubation. Anaesthesia. 2008 Sep;63(9):924-31. doi: 10.1111/j.1365-2044.2008.05525.x. Epub 2008 Jun 10. PMID 18547294
- [Background] Violet JA, Dearling JL, Green AJ, Begent RH, Pedley RB. Fractionated 131I anti-CEA radioimmunotherapy: effects on xenograft tumour growth and haematological toxicity in mice. Br J Cancer. 2008 Aug 19;99(4):632-8. doi: 10.1038/sj.bjc.6604511. PMID 18682714
- [Background] Cheville AL, Tchou J. Barriers to rehabilitation following surgery for primary breast cancer. J Surg Oncol. 2007 Apr 1;95(5):409-18. doi: 10.1002/jso.20782. PMID 17457830

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Lidocaine
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lidocaine | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (10.1) | 48.5 (7.9) | 49.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Experiencing Post Operative Nausea
Description: Nausea at any time during the post operative period for 48 hours
Time Frame: Immediate post operative to 48 hours
Measure: Number; unit: Participants
Arm/Group | Placebo | Lidocaine
Number analyzed (Participants) | 11 | 11
Participants | 11 | 11

2. Secondary Outcome: Number of Participants Experiencing Post Operative Ileus
Time Frame: 7 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Lidocaine
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

3. Primary Outcome: 24 Hour Hydromorphone
Description: Total IV hydromorphone administered during surgery to 24 hours post surgery
Time Frame: 24 hour
Measure: Mean (Standard Deviation); unit: miligrams
Arm/Group | Placebo | Lidocaine
Number analyzed (Participants) | 11 | 11
miligrams | 2.33 (1.6) | 1.5 (1.2)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Placebo | Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Lidocaine (N=11)
First degree heart block (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early because the PI left the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No